CLINICAL TRIAL: NCT02883764
Title: Cross-sectional Survey of Omega-3 Fatty Acid Blood Levels
Status: Completed | Type: Observational
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-01-031
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: eicosapentaenoic acid; EPA; docosahexaenoic acid; DHA; omega-3 index

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Employees working at DSM workplaces with an onsite Healthyroads Wellness® biometrics screening program are being offered an opportunity to have their blood fatty acids levels, especially omega-3 fatty acids [omega-3 index] measured at no charge. At some locations, participants were offered a single coupon on a 90 day supply of omega-3 capsules. Three months later, all employees at these locations are given a second opportunity to have their blood omega-3 levels [eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)] measured. The goals are to: 1) survey dietary EPA+DHA intake and omega-3 blood levels of study population, 2) determine if dietary EPA+DHA intake and omega-3 blood levels change after people have learned their omega-3 index, and 3) determine if differences in omega-3 index concentrations can be detected 3 months later between locations receiving information alone vs information+coupon.

DETAILED DESCRIPTION:
Email messages and posters announcing onsite HealthyRoads Wellness biometric screening clinics will inform ~1,800 DSM employees at 19 locations of the opportunity to participate in an omega-3 research study and have their blood omega-3 levels measured.

* Participants attending a Healthyroads Wellness® biometrics screening clinic will be invited to participate. If they agree and sign an Informed Consent form, they need to complete an Omega-3 Index Test Request form, and write their name, date of birth and collection date on the filter paper. The request form includes some dietary questions about fish/meat consumption.
* Omega-3 research participants will proceed to the biometric screening station where blood obtained from the finger stick for blood cholesterol measurements will be applied to a filter paper by a Healthyroads Wellness® professional.
* The filter paper, the Omega-3 Index Test Request, and Informed Consent form will be stapled together, packaged with all other samples obtained at that location, and shipped by DSM to a CLIA-approved laboratory.
* Within about a week of receiving the blood sample, the Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory (#43D1105229) will email the Omega-3 Index Test results directly to each participant.

Locations will be randomized such that approximately 50% of participants will receive a coupon for a discount on a 90 day supply of omega-3 capsules. These coupons will be offered to participants in order to determine rates of coupon redemption. If a coupon is offered at a biometrics screening site, a single coupon will be offered to each participant at that location. The coupon will be offered after the finger stick procedure so that it is not an incentive for participation.

Three-four months later, all employees at each location will be offered a second opportunity to have their omega-3 index measured. The filter paper, the Omega-3 Index Test Request, and Informed Consent form will be stapled together, packaged with all other samples obtained at that location, and shipped by DSM to a CLIA-approved laboratory. Based on email address, birthdate, date of collection, and gender, data will be identified as a new participant or second omega-3 index determination. This data will allow for anonymized comparison of first versus second determination of blood omega-3 index measurement to assess the impact of providing participants with information on their omega-3 status vs information + coupon.

ELIGIBILITY:
Inclusion Criteria:

* There are no exclusion criteria. These employees are 18y of age and older.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DSM offers employees to voluntarily participate in a healthyroads employee wellness program. All DSM employees working at DSM workplaces with an onsite Healthyroads Wellness® biometrics screening program will be informed by email and onsite signs of upcoming Healthyroads wellness clinics. Participants signing up for a Healthyroads Wellness clinic will be invited to participate in an omega-3 research survey.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Cross-sectional survey of omega-3 fatty acid blood levels | one day
  Single fingerstick to know blood levels of omega-3s

SECONDARY OUTCOMES:
Assessing blood levels of omega-3 fatty acids | 3 month followup
  Assessment of blood levels of omega-3 fatty acids in people 3 months after learning their omega-3 index
Assessing dietary behavior (questionnaire) | 3 month follow up
  Assessing dietary behavior in people 3 months after learning their omega-3 index

CONTACTS AND LOCATIONS:
Overall Officials: Michael I McBurney, PhD, Principal Investigator — DSM Nutritional Products, Inc.
Locations (1):
- DSM Nutritional Products, Parsippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005